CLINICAL TRIAL: NCT04288193
Title: Implementation of a Pharmacist-Driven Antipsychotic Deprescribing Initiative in the Program of All-inclusive Care for the Elderly (PACE) Setting: A Pilot Study
Brief Title: Implementation of a Pharmacist-Driven Antipsychotic Deprescribing Initiative in the PACE Setting: A Pilot Study
Status: Withdrawn | Type: Observational
Why Stopped: Change in personnel, unable to begin project.
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: RPH-APDP-001
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia; Insomnia
Keywords: sleep; antipsychotic; bpsd; deprescribing
MeSH Terms: conditions — Behavior; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trinity Health LIFE New Jersey PACE: Participants enrolled in Trinity Health LIFE New Jersey PACE facility who received an antipsychotic medication for the treatment of BPSD or insomnia
  Interventions: Drug: Recommendation to Deprescribe

INTERVENTIONS:
Drug: Recommendation to Deprescribe — Recommendation to Deprescribe

SUMMARY:
The aim of this pilot study is to determine the feasibility of implementing an antipsychotic deprescribing initiative that is driven by pharmacists working collaboratively with the Program of All-inclusive Care for the Elderly (PACE) interdisciplinary team.

DETAILED DESCRIPTION:
No individual antipsychotic has been approved by the U.S. Food and Drug Administration (FDA) for treating insomnia or behavioral and psychological symptoms of dementia (BPSD). Despite these medications being associated with significant harms, a considerable portion of older adults are prescribed antipsychotics for treatment of insomnia or BPSD. The aim of this study is to determine the feasibility of a pharmacist-driven antipsychotic deprescribing initiative in a community-based practice setting known as Program of All-inclusive Care for the Elderly (PACE). Our primary objective is to assess and describe the implementation process, including barriers and enablers to implementation. Our secondary objectives are to quantify and describe changes in antipsychotic prescribing following implementation; evaluate and report on antipsychotic re-initiations or changes in dosing; and evaluate and report on adverse drug withdrawal events (ADWEs) following antipsychotic deprescribing.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled in a PACE organization during the implementation time period;
* PACE organization contractually receiving pharmacy services from CareKinesis during the implementation time period; and,
* Participant's prescriber determines that the participant could potentially benefit from deprescribing the antipsychotic.

Exclusion Criteria:

* A diagnosis of bipolar disorder, schizophrenia, schizo-affective disorder, acute delirium, Tourette's syndrome, tic disorders, autism, intellectual disability, developmental delay, obsessive-compulsive disorder, alcoholism, cocaine abuse, Parkinson's disease psychosis, or major depressive disorder for which the antipsychotic is specifically prescribed as adjunctive treatment;
* Participant's prescriber determines that the participant would likely not benefit or could be harmed from deprescribing the antipsychotic; and,
* Participant, or healthcare decision-maker on behalf of the participant (e.g., caregiver) refuses to participate in the deprescribing initiative.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Program of All-inclusive Care for the Elderly (PACE) is a Medicare-Medicaid program that provides comprehensive medical and supportive services to individuals >55 years of age who are certified by their state as needing nursing home care but are able to live safely in the community through PACE, as an alternative to institutionalization.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-05-18 (Estimated); Study Completion 2022-05-18 (Estimated)

PRIMARY OUTCOMES:
Identify barriers and enablers to implementation of antipsychotic deprescribing initiative. | Three months
  Qualitative

SECONDARY OUTCOMES:
Implement changes in antipsychotic prescribing to patients in the PACE population. | Three months
  Quantitative and Qualitative
Measure the number of antipsychotic re-initiations in the PACE population. | Three months
  Quantitative
Measure changes in antipsychotic dosing for the PACE population. | Three months
  Quantitative
Identify the number of adverse drug withdrawal events (ADWEs) in the PACE population. | Three months
  Quantitative and Qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, PhD, Principal Investigator — Tabula Rasa HealthCare; Anna Furman, PharmD, Principal Investigator — Tabula Rasa HealthCare; Adriana Matos, PharmD, Principal Investigator — Tabula Rasa HealthCare; Nishita Amin, PharmD, Principal Investigator — Tabula Rasa HealthCare; Briana Skalski, PharmD, Principal Investigator — Tabula Rasa HealthCare; Sweilem Al Rihani, PhD, PharmD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Trinity Health LIFE, New Jersey, Pennsauken, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bain KT, Holmes HM, Beers MH, Maio V, Handler SM, Pauker SG. Discontinuing medications: a novel approach for revising the prescribing stage of the medication-use process. J Am Geriatr Soc. 2008 Oct;56(10):1946-52. doi: 10.1111/j.1532-5415.2008.01916.x. Epub 2008 Sep 2. PMID 18771457
- [Background] Jeste DV, Blazer D, Casey D, Meeks T, Salzman C, Schneider L, Tariot P, Yaffe K. ACNP White Paper: update on use of antipsychotic drugs in elderly persons with dementia. Neuropsychopharmacology. 2008 Apr;33(5):957-70. doi: 10.1038/sj.npp.1301492. Epub 2007 Jul 18. PMID 17637610
- [Background] Feng Z, Hirdes JP, Smith TF, Finne-Soveri H, Chi I, Du Pasquier JN, Gilgen R, Ikegami N, Mor V. Use of physical restraints and antipsychotic medications in nursing homes: a cross-national study. Int J Geriatr Psychiatry. 2009 Oct;24(10):1110-8. doi: 10.1002/gps.2232. PMID 19280680
- [Background] Yan J. FDA extends black-box warning to all antipsychotics. Psychiatric News. 2008;43:1-27.
- [Background] US Government Accountability Office. Antipsychotic drug use: HHS has initiatives to reduce use among older adults in nursing homes, but should expand efforts to other settings. Washington, DC: US Government Accountability Office; 2015.
- [Background] U.S. Food and Drug Administration. Information for healthcare professionals: conventional antipsychotics. Silver Spring, MD: Center for Drug Evaluation and Research. 2008.
- [Background] Wetzels RB, Zuidema SU, de Jonghe JF, Verhey FR, Koopmans RT. Prescribing pattern of psychotropic drugs in nursing home residents with dementia. Int Psychogeriatr. 2011 Oct;23(8):1249-59. doi: 10.1017/S1041610211000755. Epub 2011 Jun 20. PMID 21682938
- [Background] U.S. Food and Drug Administration. Public health advisory:deaths with antipsychotics in elderly patients with behavioral disturbances. Silver Spring, MD: Center for Drug Evaluation and Research. 2005.